CLINICAL TRIAL: NCT02770560
Title: Efficacy of Urokinase Containing Locking Solutions for Thrombotic Dysfunction of Tunneled Cuffed Catheters : a Single-center Retrospective Study
Brief Title: Efficacy of Urokinase Containing Locking Solutions for Thrombotic Dysfunction of Tunneled Hemodialysis Catheters
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2015-12-24; First posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2015-12

CONDITIONS: Kidney Failure, Chronic; Vascular Access Devices
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic hemodialysis patients with a tunneled cuffed catheter: In case of thrombotic dysfunction of the dialysis catheter : administration of Urokinase (100 000 units in total) as locking solution in the dead space of the catheter lumen, interdialytic (between two dialysis sessions) or intradialytic (during the dialysis in case of complete obstruction of the dialysis catheter)
  Interventions: Device: Urokinase locking solution

INTERVENTIONS:
Device: Urokinase locking solution — On basis of the prescription : one single administration of thrombolytic locking solution versus multiple administrations (during 3 consecutive dialysis sessions)
  Other Names: Actosolv

SUMMARY:
Thrombotic dysfunction is a common complication of tunneled cuffed catheters (TCC) leading to inadequate dialysis dose, need to catheter replacement with as consequence progressive exclusion of vascular sites. Thrombolytic agent can be used as therapeutic locking solution to dissolve the clotting formed in of around the catheter lumen. There are few studies on the optimal approach of TCC-related thrombosis with thrombolytic containing locking solution (dose, number of administrations, timing of administration - intra or interdialytic use). The primary objective of this retrospective study was to compare the efficacy of inter versus intradialytic Urokinase containing locking solution on restoration of the TCC blood flow. The investigators also assess the question of multiple administrations of Urokinase are more efficient than one single administration

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patients over 18 years old, receiving hemodialysis between 1st May 2010 and 31st October 2014 via a tunneled cuffed catheter at the Hemodialysis Unit of Universitair Ziekenhuis Brussel Hospital.

Exclusion Criteria:

* Patients younger than 18 years old
* Patients with a temporary dialysis catheter
* Patients who never received a tunneled hemodialysis catheter in this period
* Patients who didn't have a medical file at the Universitair Ziekenhuis Brussel Hospital

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Incident and prevalent patients on hemodialysis, more than 18y old, receiving dialysis via a tunneled cuffed catheter between 1st May 2010 and 31st October 2014.
Sampling Method: Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2010-05; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in catheter blood flow (expressed in ml/min) after Urokinase-containing locking solution | up to 54 months
  Comparison of catheter blood flow measurement before and after Urokinase locking solution administration according to the type of Urokinase prescription (inter- versus intra-dialytic use, one- single versus multiple administrations)
Change of pump pressures (expressed in mmHg) after Urokinase-containing locking solution | up to 54 months
  Comparison of pump pressures measurement before and after Urokinase locking solution administration according to the type of prescription of Urokinase containing locking solution (inter versus intra-dialytic, one single use versus multiple administrations)

CONTACTS AND LOCATIONS:
Overall Officials: Florence Bonkain, M.D., Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No